CLINICAL TRIAL: NCT00745784
Title: Lost to Cancer: Prolonged Grief in Young Bereaved Spouses and Partners
Brief Title: Prolonged Grief in Young Bereaved Spouses and Partners
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Calvary Hospital, Bronx, NY (Other)
Responsible Party: Andrew Roth, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 08-100
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Grief
Keywords: Young Bereaved Spouses
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Young spouses/domestic partners (20-49 years old) of cancer patients who have died from cancer.
  Interventions: Behavioral: in-person or telephone interview

INTERVENTIONS:
Behavioral: in-person or telephone interview — Participants will be administered one battery of questionnaires that should take 50- 55 minutes, which may be broken down into two or more segments if necessary. They may choose to have these questionnaires administered to them in person at the hospital, in person at their home, or via telephone by a trained master's level research assistant.

SUMMARY:
The purpose of the research is to learn more about the experience of grief in young bereaved spouses/partners. Recent research has shown that young bereaved spouses/partners experience grief uniquely from other age groups, but it is still unclear how certain factors affect the experience of grief. The investigators research team is interested in studying how the psychological factors of trauma, personality, and meaning of the loss affect grief reactions in young spouses/partners after the loss of a spouse to cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 20 years old and no older than 49 years and 11 months old.
* Participants must have lost a spouse/domestic partner to cancer 6 months to 3 years earlier.
* Participants must be able to give informed consent.
* Participants must be able to comprehend English to complete study assessments.

Exclusion Criteria:

* Major psychopathology or cognitive impairment likely in the judgment of the research staff to interfere with the participation or completion of the protocol.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Only spouses/partners of deceased Calvary and Memorial Sloan Kettering patients will be assessed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To determine the rate and levels of prolonged grief in young bereaved spouses/partners of cancer patients | conclusion of the study

SECONDARY OUTCOMES:
To determine associations among prolonged grief, personality characteristics , previous trauma, & subjective meanings of the loss to the bereaved spouse in young bereaved spouses/partners of cancer | conclusion of the study
To evaluate whether unique themes emerge among those reporting prolonged grief | conclusion of the study
To evaluate whether unique themes emerge among those reporting obsessive and histrionic personality traits | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Schacter, PhD, Principal Investigator — Calvary Hospital, Bronx, NY
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Calavery Hospital, The Bronx, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org